CLINICAL TRIAL: NCT02576132
Title: Pupillometry for Pain Assessment in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Other Study IDs: Vola-ICU
Record Dates: First submitted 2015-10-09; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was part of a quality improvement project at the Department of Anesthesiology and Intensive Care Medicine, Charité - Universitaetsmedizin Berlin.

Being in pain is reported to be one of the most important stressors in critically ill patients and worsens outcome. The evaluation of pain using validated scores in patients who are able to self-report significantly improves the quality of analgesic therapy and health related outcomes in intensive care patients.

However, behavioral pain score that are used in sedated or delirious patients, often underestimate the severity of pain.

The primary aim of this study is to investigate if measurement of the pupillary light reflex Amplitude correlates with the results of pain assessment using validated pain scores in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* aged 18 years or older
* patients with an expected intensive care unit length of stay of of at least 48 hours.

Exclusion Criteria:

* not German speaking
* traumatic brain injury
* stroke
* increased intracranial pressure
* ocular disease or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients, aged 18 years or older with an expected intensive care unit length of stay of of at least 48 hours.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient of pupillary light reflex amplitude and pain score | Participants will be followed up to 6 days during their intensive care unit stay
  Pain is measured by Numeric Rating Scale - Visualised or Behavioural Pain Scale or Behavioral Pain Scale - Non Intubated and pupillary light reflex amplitude is measured by pupillometry

SECONDARY OUTCOMES:
Minimal pupil size [mm] | Participants will be followed up to 6 days during their intensive care unit stay
Maximal pupil size [mm] | Participants will be followed up to 6 days during their intensive care unit stay
Contraction speed of pupil [mm/s] | Participants will be followed up to 6 days during their intensive care unit stay
Latency of pupil [ms] | Participants will be followed up to 6 days during their intensive care unit stay
Pupillary light reflex [%] | Participants will be followed up to 6 days during their intensive care unit stay
Richmond Agitation Sedation Scale (RASS) | Participants will be followed up to 6 days during their intensive care unit stay
Glasgow Coma Scale (GCS) | Participants will be followed up to 6 days during their intensive care unit stay
Delirium | Participants will be followed up to 6 days during their intensive care unit stay
  Delirium is measured by the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)
Duration of mechanical ventilation (hours) | Participants will be followed up during their intensive care unit stay, an average of 25 days
Intensive care unit length of stay (days) | Participants will be followed up during their intensive care unit stay, an average of 25 days
Hospital length of stay (days) | Participants will be followed up during their hospital length of stay, an average of 5 weeks
Hospital mortality (days) | Participants will be followed up during their hospital length of stay, an average of 5 weeks
Discharge to home [%] | Participants will be followed up during their hospital length of stay, an average of 5 weeks
Morbidity Scores | Participants will be followed up during their intensive care unit stay, an average of 25 days
Amount of administered drugs | Participants will be followed up to 6 days during their intensive care unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Charité - Univeritätsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine, Berlin, State of Berlin, Germany